CLINICAL TRIAL: NCT01116297
Title: Tissue Oxygenation Measurements During Plastic Surgery Using Spatially Modulated Light (S-FLARE)
Brief Title: Tissue Oxygenation Measurements With Modulated Light (S-FLARE)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, John V. Frangioni, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009-P000384 BIDMC
Record Dates: First submitted 2010-02-03; First posted 2010-05-04 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Breast Cancer
Keywords: breast reconstruction; breast cancer; near infrared imaging
MeSH Terms: conditions — Breast Neoplasms | interventions — Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imaging with S-FLARE imaging system (Experimental): 3 patients to be imaged by S-FLARE imaging system.
  Interventions: Device: Imaging with S-FLARE imaging system

INTERVENTIONS:
Device: Imaging with S-FLARE imaging system — Tissue oxygenation measurements during plastic surgery using the S-FLARE system.

SUMMARY:
To perform a pilot study of the S-FLARE imaging system, which uses low levels of safe, invisible, near-infrared light to measure tissue oxygenation during breast reconstructive surgery and to compare S-FLARE measurements to the gold standard, FDA-approved, the ViOptix optical probe.

DETAILED DESCRIPTION:
This pilot study will enroll three patients who have chosen to proceed with deep inferior epigastric perforator (DIEP) flap breast reconstruction. This type of reconstruction uses skin and fat from the abdomen to reconstruct a new breast shape. The construct is vascularized through perforating arteries and veins that provide a blood supply to this tissue.

Current techniques to evaluate vessel selection rely on a handheld Doppler used for confirmation of blood flow and perfusion; however, this modality is limited as it only assesses a specific point within the flap.

The S-FLARE imaging system will be used to visualize vascularization in the DIEP flaps, and this study will compare measurements by the S-FLARE imaging system and the standard-of-care ViOptix point probe.

ELIGIBILITY:
Inclusion Criteria:

* Women or men above the age of 21 who are undergoing unilateral breast reconstruction after mastectomy.
* Women of childbearing age must have a negative pregnancy test as confirmed by anesthesiologist.

Exclusion Criteria:

* BMI > 30.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Optimization of Ergonomics and Functioning of the S-FLARE Imaging System during Breast Reconstructive Surgery | 10 minute imaging procedure
  Due to patient-to-patient anatomic variation, the vascular perfusion to the skin in DIEP flaps is unpredictable and of great concern to the surgeon planning the flap design. We propose a method of imaging tissue oxygenation within a DIEP flap base on the use of invisible near-infrared light.
  This pilot study is a comparison study of oxygenation measurements taken by the ViOptix optical probe as the standard of care and the S-FLARE imaging system, with the intention of optimizing the ergonomics and functionality of the S-FLARE imaging system for use during breast reconstructive surgery.

CONTACTS AND LOCATIONS:
Overall Officials: John V. Frangioni, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- See also: Website of the study principal investigator with detailed information about related work. — http://www.frangionilab.org